CLINICAL TRIAL: NCT05597241
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Dose and Multiple Ascending Dose, Single Center Phase1 Study of Safety, Tolerability, Pharmacokinetics, and Electroencephalography of Intravenous GATE-202 in Healthy Volunteers
Brief Title: Multiple Ascending Dose and Electroencephalography Trial of GATE-202 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndeio Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GATE-202-C-101
Record Dates: First submitted 2022-10-21; First posted 2022-10-28 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-10

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; single ascending dose; multiple ascending dose; pharmacokinetics; EEG
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1, Apimostinel (Experimental): Apimostinel, 25 mg IV single dose
  Interventions: Drug: apimostinel
- Cohort 1, Placebo (Placebo Comparator): Placebo, IV single Dose
  Interventions: Drug: Placebo
- Cohort 2, Apimostinel, 1 mg IV 8 consecutive daily doses (Experimental): Apimostinel, 1 mg IV 8 consecutive daily doses
  Interventions: Drug: apimostinel
- Cohort 2, Placebo IV 8 consecutive daily doses (Placebo Comparator): Placebo IV 8 consecutive daily doses
  Interventions: Drug: Placebo
- Cohort 3, Apimostinel, 5 mg IV 8 consecutive daily doses (Experimental): Apimostinel, 5 mg IV 8 consecutive daily doses
  Interventions: Drug: apimostinel
- Cohort 3, Placebo 8 consecutive daily doses (Placebo Comparator): Placebo IV 8 consecutive daily doses
  Interventions: Drug: Placebo
- Cohort 4, Apimostinel, 10 mg IV 8 consecutive daily doses (Experimental): Apimostinel, 10 mg IV 8 consecutive daily doses
  Interventions: Drug: apimostinel
- Cohort 4, Placebo 8 consecutive daily doses (Placebo Comparator): Placebo IV 8 consecutive daily doses
  Interventions: Drug: Placebo
- Cohort 5, Apimostinel, 25 mg IV, 8 consecutive daily doses (Experimental): Apimostinel, 25 mg IV 8 consecutive daily doses
  Interventions: Drug: apimostinel
- Cohort 5, Placebo IV 8 consecutive daily doses (Placebo Comparator): Placebo IV 8 consecutive daily doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: apimostinel — N-methyl-D-aspartate (NMDA) receptor modulator
  Other Names: GATE-202
  Arms: Cohort 1, Apimostinel; Cohort 2, Apimostinel, 1 mg IV 8 consecutive daily doses; Cohort 3, Apimostinel, 5 mg IV 8 consecutive daily doses; Cohort 4, Apimostinel, 10 mg IV 8 consecutive daily doses; Cohort 5, Apimostinel, 25 mg IV, 8 consecutive daily doses
Drug: Placebo — Placebo
  Arms: Cohort 1, Placebo; Cohort 2, Placebo IV 8 consecutive daily doses; Cohort 3, Placebo 8 consecutive daily doses; Cohort 4, Placebo 8 consecutive daily doses; Cohort 5, Placebo IV 8 consecutive daily doses

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and EEG pharmacodynamics of single and multiple ascending doses of apimostinel in normal human volunteers

DETAILED DESCRIPTION:
Single ascending dose (SAD), multiple ascending dose (MAD), double-blind placebo-controlled study in normal human volunteers.

Subjects will receive a single 25 mg IV dose of apimostinel or matching placebo, or 8 consecutive days of 1, 5, 10, or 25 mg IV or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a healthy volunteer who is able to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.
2. Subject must be 18 to 55 (inclusive) years of age, at the time of signing the informed consent.
3. Subject has a BMI between 18.5 kg/m2 and 30 kg/m2 (inclusive), with a minimum body weight of 50 kg.
4. Subject is male or female.
5. Females are eligible to participate if not pregnant, not breastfeeding, and at least one of the following conditions applies:

   * Surgically sterile or at least 2 years menopausal, confirmed by follicle-stimulating hormone (FSH) at Screening, or,
   * If women of childbearing potential (WOCBP), subject must use an acceptable method of birth control from date of Screening to at least 30 days after the last dose of study intervention and must have a documented negative blood or urine pregnancy test within 24 hours prior to dosing (SAD cohort) or within 48 hours prior to dosing (MAD cohorts). If reported sterile or postmenopausal, will be confirmed by FSH.
6. Male subject must meet one of the following:

   * Surgically sterile
   * If not surgically sterile, then use of an acceptable form of contraception as detailed in Appendix 4 from the time of randomization through 28 days following the last dose of study intervention. Male subjects or male partners of female subjects are recommended to not donate sperm from Screening (Visit 1) until 28 calendar days after the last dose of study intervention. Male subjects are strongly advised to inform female partners of the need for them to use acceptable birth control methods during this time period.
7. Clinical laboratory values <2 times the upper limit of normal or deemed not clinically significant by the Investigator at Screening and Admission Day.

Exclusion Criteria:

1. Type I or Type II diabetes mellitus.
2. Malignancy in the last 5 years, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
3. History of allergy or sensitivity, or intolerance to N-methyl-D-aspartate (NMDA) receptor ligands including ketamine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone.
4. Psychiatric disease including major depressive disorder, bipolar disorder, anxiety, or schizophrenia, or other medical condition that, in the opinion of the Investigator, would interfere with the evaluation of study intervention safety.
5. Any personal or family history of seizure (including febrile seizures) or diagnosis of epilepsy or episode of unexplained loss of consciousness.
6. Any history of neurological or other medical conditions which in the opinion of the Investigator has the potential to reduce seizure threshold, e.g., history of head concussion, traumatic brain injury, taking any medications that may reduce seizure threshold, developmental abnormalities in the brain, or metabolic causes, including electrolyte abnormalities such as hyponatremia.
7. Subject has a history of excessive bleeding after invasive procedures or surgery or known coagulation or platelet abnormality or has been on any blood thinner or medication affecting platelet function, such as aspirin, nonsteroidal antiinflammatory medications, corticosteroids (except topical) or warfarin within the 7 days prior to enrollment or has known allergy to any anesthetic agent that may be used for the lumbar catheterization.
8. Subject has a history of infection that required IV antibiotics within the 45 days or oral antibiotics within 30 days prior to enrollment, and, at the time of clinic admission, be febrile or have signs/symptoms consistent with an infection.
9. Subject has a history of or physical examination evidence of a lumbar spine abnormality that may preclude placement of a spinal catheter, presence of intraspinal shunt devices (e.g., ventriculoperitoneal shunt), or history of elevated intracranial pressure, normal pressure hydrocephalus, or other neurological condition that in the opinion of the Investigator precludes safe study participation. A lumbar X-ray that excludes spine abnormalities must have been taken within the past 12 months and made available or the subject must agree to have one taken as part of the qualification.
10. In the opinion of the Investigator, the Safety Monitor, or the Sponsor Study Monitor, has a history of severe renal or hepatic impairment, severe active hepatic disease, or other clinically significant medical condition that may preclude safe study participation.
11. Subject who has clinical signs and symptoms consistent with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); e.g., fever, dry cough, dyspnea, sore throat, fatigue, or positive SARS-CoV-2 test result within 14 days prior to the Screening Visit or at admission.
12. Subject who had a severe course of SARS-CoV-2 (extracorporeal membrane oxygenation, mechanically ventilated).
13. Currently taking prescription or over-the-counter medications including herbal therapies, within 14 days of enrollment into the study.
14. Received another investigational drug or device within 30 days or 5 half-lives, whichever is longer prior to enrollment in this study (defined as the time of admission; Day -2 for MAD and Day -1 for SAD).
15. Previously randomized in this study.
16. Has a positive test for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or human immunodeficiency virus (HIV) at Screening or has been previously treated for hepatitis B, hepatitis C, or HIV infection.
17. For Cohorts 2-5, evidence of hearing loss that cannot be compensated for in the event related potential (ERP) tests, assessed by audiologic examination.
18. Evidence of alcohol abuse, defined as regular consumption of alcohol within 6 months prior to screening defined as > 7 drinks/week for females and > 14 drinks/week for males where 1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor. Use of illicit substances and recreational drug use (such as marijuana) within 3 months prior to the Screening Visit is also prohibited.
19. Current abuse of illicit substances, using the Diagnostic and Statistical Manual V definition of substance use disorder.
20. Has a positive urine screen for drugs of abuse (see Table 10 1) at Screening and admission day (Day -2 for MAD and Day -1 for SAD).
21. Currently pregnant, planning to become pregnant during the course of the study, or nursing mother.
22. At Screening, if the Columbia-Suicide Severity Rating Scale (C-SSRS) responses ("yes" answers to item 4 or 5) indicate that the subject may have experienced suicidal ideation associated with actual intent or plan within 12 months of Screening, may have had a history of suicidal behavior within the past 10 years, or had any lifetime history of recurrent suicidal behavior, the subject will be excluded from participation in the study.
23. Previous cerebrospinal fluid (CSF) collection within 30 days prior to admission to the clinical research unit.
24. Impaired function (glomerular filtration rate <60 mL/min) by the chronic kidney disease-Epidemiological Collaboration (CKD-EPI Creatinine) calculation method. Can be repeated once during Screening and once during admission.
25. Elevated systolic blood pressure (>140 mmHg) or diastolic blood pressure (>90 mmHg) and/or increased corrected QT interval (QTc) (>450 msec for men or >470 msec for women) or additional risk factors for Torsades de Pointes including heart failure, hypokalemia, or family history of Long QT Syndrome at Screening or Admission Day. Can be repeated once during Screening and once during admission.
26. Has donated blood (≥500 mL) or blood products within 6 weeks (42 days) prior to admission.
27. Subject is deaf or has hearing loss of more than 25 decibels (dB) in one or both ears.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | 36 days
  Number of Participants with Treatment-Emergent Adverse Events Through Study Completion

SECONDARY OUTCOMES:
Pharmacokinetics - Maximum Plasma Concentration | 72 hours
  Maximum observed plasma concentration after a single dose or after 8 doses

OTHER OUTCOMES:
EEG - Power | 6 hours
  Changes in EEG band power
Event related potential (ERP) | 6 hours
  P300

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Burch, MD PhD, Principal Investigator — Syndeio Biosciences, Inc
Locations (1):
- Woodland Research Northwest, Rogers, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No